CLINICAL TRIAL: NCT04340622
Title: A Project to Test The Efficacy And Safety Of An Innovative Treatment Of Opiate Use Disorders
Brief Title: Efficacy And Safety Of An Innovative Treatment Of Opiate Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MindLight, LLC (Industry)
Collaborators: Mclean Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R43DA050358 (NIH); 1R43DA050358-01 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2020-04-09 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: 20 participants will receive twice a week active treatment for 4-weeks of a 4-minute near-infrared light treatment through the forehead to a brain hemisphere and 20 will receive a sham treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The sham is created by putting a piece of aluminum foil over the light-emitting diode. It will be placed there or not placed there by a 3rd party so that neither the participant nor the outcomes assessor will know the condition of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reduction in opioid cravings and use (Active Comparator): These participants will receive twice-weekly transcranial photobiomodulation with and 810 nm LED for 4 min for a delivery to the brain of 2.1 J/cm2. The treatment will last 4 weeks. We anticipate a 60% reduction in opioid cravings in this group. We anticipate a reduction of at least 1.6 days of use per week on average.
  Interventions: Device: supra-luminous LED
- Small reduction in opioid cravings and use (Placebo Comparator): Sham condition.
  Interventions: Device: Sham

INTERVENTIONS:
Device: supra-luminous LED — 810 nm light-emitting diode for the delivery of 2.1 J/cm2 to the brain.
  Other Names: unilateral trancranial photobiomodulation, near-infrared mode
  Arms: Reduction in opioid cravings and use
Device: Sham — Light-emitting diode covered with aluminium foil
  Arms: Small reduction in opioid cravings and use

SUMMARY:
Investigators will test, for safety and efficacy, a novel treatment for opiate addiction that applies a 4-minute treatment of intense near infra-red light to stimulate a side of the brain that the investigators determine to be healthier, more mature, and less traumatized. Investigators will compare an active and a sham treatment given twice weekly for 4-weeks. Investigators hope this will lead to a significant weapon in the battle against the opioid epidemic as well as lead to psychological and physiological insights into possible relations among trauma, cerebral laterality, and addiction.

DETAILED DESCRIPTION:
This project is to demonstrate that a novel treatment for opiate addiction is safe and far superior to a sham comparison treatment. The treatment is hoped to significantly aid in the battle against the opioid epidemic that is ravaging much of the country and the world. The treatment consists of using a 4-minute application of transcranial photobiomodulation, near infra-red mode, through a supra-luminous LED, to one side of the forehead over the brain hemisphere that we determine (through a proprietary test) to have a more positive emotional valence. Based on preliminary data, we anticipate that the treatment will be very effective in reducing drug cravings, anxiety, and depression as well as in reducing relapses. Aim I will offer twice-weekly treatments to two groups, active and sham, for 4-weeks and will look specifically for differences in opioid cravings, anxiety, depression, and opioid use. The investigators will evaluate participants weekly for safety and efficacy for 3-weeks post-treatment. In Aim II a highly-regarded product engineer will work with the company to design a marketable product that may have patentable elements.

ELIGIBILITY:
Inclusion Criteria:

* all patients must between the ages of 18 and 70
* meet criterion for a history of Opioid Use Disorder (OUD) on a Diagnostic Interview.
* have opioid cravings
* Enrollment will be made without regard to gender or ethnicity.
* Patients who are receiving treatment for OUD or other psychiatric disorders, either psychological or pharmacological treatments, may continue their treatment during the time of the study but will be asked to try not to alter their treatment from the onset of the experiment until its conclusion. The statistical analysis will include covariates for doses of buprenorphine and methadone and use of non-prescribed opioids

Exclusion Criteria:

* past history of a psychotic disorder (including schizophrenia or schizoaffective disorder)
* history of violent behavior
* history of a past suicide gesture or attempt, a history of current suicidal ideation, *history of a neurological condition (e.g. epilepsy, traumatic brain injury, stroke), *pregnancy
* current acute or chronic medical condition requiring a medication that has psychological side-effects.
* impaired decision-making capacity in the judgment of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Opioid Craving Scale | One year
  a published 3 question scale of opioid cravings. Each question asks the patient to rate his opioid cravings at the present time from 0 (none) to 9 (extreme). We use the average of the scores of the 3 questions. A low score is best.
Change in Opioid drug use | One year
  TimeLine FollowBack method, measures the daily amount of opioid drug use (mg's of pills or grams used) for the period between observations.

SECONDARY OUTCOMES:
Change in Patient reports of opioid use by TimeLine FollowBack method | One year
  patient reports supported by urine drug screens and a drug hair test at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Schiffer, MD, Principal Investigator — MindLight, LLC; Martin Teicher, MD, PhD, Principal Investigator — McLean Hospital and Harvard Medical School
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - MindLight, LLC, Newton Highlands, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Without any identifying participant information, study data may be shared at the investigator's discretion.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: upon completion of the study
Access Criteria: Investigators will not share any individual participant identifying data. Each participant will be given a participant number and this number will be shared with the participant's data. All participant data will be shared but without any participant, personal identifying data.

REFERENCES:
- [Derived] Schiffer F, Khan A, Bolger E, Flynn E, Seltzer WP, Teicher MH. An Effective and Safe Novel Treatment of Opioid Use Disorder: Unilateral Transcranial Photobiomodulation. Front Psychiatry. 2021 Aug 10;12:713686. doi: 10.3389/fpsyt.2021.713686. eCollection 2021. PMID 34447323